CLINICAL TRIAL: NCT02561442
Title: A Single-Dose, Randomized, Three-way, Partially Blinded Crossover Study to Compare the Pharmacokinetics and Bioavailability of Ceftriaxone Administered as a 1 Gram Intravenous Infusion, a 1 Gram Subcutaneous Infusion and a 2 Gram Subcutaneous Infusion in Healthy Adult Subjects
Brief Title: Crossover Study to Compare the Pharmacokinetics of Subcutaneous and Intravenous Ceftriaxone Administration
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: scPharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: scP-02-001
Record Dates: First submitted 2015-09-24; First posted 2015-09-28 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Pharmacokinetics in Healthy Adults
MeSH Terms: interventions — Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IV ceftriaxone (0.5hr) 1 gm (Active Comparator): ceftriaxone for injection, (total dose = 1.0 g) administered IV over 30 minutes via infusion pump (Open Label)
  Interventions: Drug: ceftriaxone
- subcutaneous ceftriaxone, (2hr), 1 gm (Experimental): ceftriaxone for injection, (total dose = 1.0 g) administered subcutaneous over 2 hours (Blinded).
  Interventions: Drug: ceftriaxone
- subcutaneous ceftriaxone, (2 hr), 2 gm (Experimental): ceftriaxone for injection, (total dose = 2.0 g) administered subcutaneous over 2 hours (Blinded).
  Interventions: Drug: ceftriaxone

INTERVENTIONS:
Drug: ceftriaxone

SUMMARY:
The proposed study aims to assess the time above MIC (4 mg/mL), and the pharmacokinetics/pharmacodynamics and bioavailability of 1 g ceftriaxone administered by constant rate subcutaneous infusion over 2 hours compared with 1 g of ceftriaxone administered as a constant IV infusion over 0.5 hours. In addition, the study will compare the results obtained after 1 g ceftriaxone intravenous or subcutaneous administration with 2 g ceftriaxone administered subcutaneously

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
2. Male and female subjects between 18 and 65 years of age inclusive.
3. Subjects must have body weight of 45.5 to 105 kg inclusive and body mass index (BMI) ≤34 kg/m2.
4. Females will be non-pregnant, non-lactating, and either post-menopausal for at least 1 year, surgically sterile (e.g., tubal ligation, hysterectomy) for at least 90 days, or agree, from the time of signing the informed consent or 14 days prior to Baseline until Follow-up, to use TWO (2) of the following forms of contraception: a IUD with spermicide, female condom with spermicide, contraceptive sponge with spermicide, an intravaginal system, diaphragm with spermicide, cervical cap with spermicide, a male sexual partner who agrees to use a male condom with spermicide, a sterile sexual partner, OR abstinence. For all females, a pregnancy test result must be negative at Screening and Baseline/Day 0
5. Males agree from the time of Baseline/Day 0 until Follow-up, to use TWO (2) forms of contraception: ONE must be a male condom with spermicide; the second may be ONE of the following: his female partner uses either an IUD with spermicide, female condom with spermicide, contraceptive sponge with spermicide, an intravaginal system, diaphragm with spermicide, cervical cap with spermicide, oral contraceptives; OR abstinence
6. Subject has normal (or abnormal and clinically insignificant) laboratory values at screening.
7. Subject is medically normal with no significant abnormal findings at the Baseline physical examination.
8. Subjects must have Baseline values of the following laboratory tests as specified:

   * AST, ALT, alkaline phosphatase (ALP), total bilirubin, and creatinine <1.1 ULN
   * Platelet count >100 X 103/µL
   * Neutrophil count >1.0 X 103/µL
9. Subject has the ability to understand the requirements of the study and is willing to comply with all study procedures.
10. Subject has not consumed and agrees to abstain from taking any vitamin or dietary supplements or non-prescription drugs (except as authorized by the Investigator and Medical Monitor) for 3 days prior to CRU admission through Follow-Up, with the exception of oral contraceptives.
11. Subject has not consumed and agrees to abstain from taking any prescription drugs (except as authorized by the Investigator and Medical Monitor) during the 14 days prior to CRU admission through Follow-Up.
12. Subject has not consumed and agrees to abstain from consuming grapefruit, grapefruit juice, or juices containing grapefruit, or Seville oranges during the 3 days prior to CRU admission through Follow-Up.
13. Subject agrees to abstain from using alcohol from 48 hours prior to Screening and CRU admission through CRU discharge for each period.

Exclusion Criteria:

1. Evidence of or history of clinically significant oncologic, pulmonary, hepatic, gastrointestinal, cardiovascular, hematologic, metabolic, neurological, immunologic, nephrologic, endocrine, or psychiatric disease, or current clinically significant infection.
2. History of chronic skin conditions requiring medical therapy.
3. Clinically significant abnormalities at Screening or Baseline in safety laboratory tests.
4. Corrected QT interval (QTc) greater than 450 msec for males and 470 msec for females as corrected by the Fridericia formula.
5. Major surgery within 30 days prior to Screening.
6. Administration of an investigational drug or implantation of investigational device, or participation in another trial, within 30 days prior to Screening.
7. Any surgical or medical condition which in the opinion of the investigator may interfere with participation in the study or which may affect the outcome of the study.
8. Positive test for hepatitis B, hepatitis C, or HIV at Screening.
9. Positive urine drug screen at Screening or Baseline.
10. Tobacco users (includes users who stopped smoking £90 days prior to the screening evaluation). [Note: "Tobacco use" includes smoking and the use of snuff and chewing tobacco, and other nicotine or nicotine containing products.]
11. History of alcohol abuse within 6 months prior to screening, as determined by the Investigator.
12. Consumed alcohol within 48 hours of Screening or each CRU admission or have a positive alcohol test at Screening or any admission to the CRU.
13. Known allergy cephalosporin class of antibiotics or penicillin.
14. Female subject who is pregnant or lactating.
15. Donation of greater than 100 mL of either whole blood or plasma within 30 days prior to study drug administration.
16. Subjects with hemoglobin (Hb) ≤10.5 g/dL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration | 48 hours
  Cmax, observed by inspection of individual study participant plasma concentration time plots.
Time of observed maximum plasma concentration | 48 hours
  Tmax, obtained directly from the observed concentration-time data
Area under the plasma concentration-time curve | 48 hours
  AUClast: AUC from time 0 to the last measureable non-zero concentration, calculated by a combination of linear and logarithmic trapezoidal methods
Area under the concentration time curve, extrapolated to infinity | 48 hours
  AUCinf: Area under the concentration time curve from time 0 extrapolated to infinity, calculated as AUClast + Clast/λz
Terminal phase elimination rate constant | 48 hours
  Terminal phase elimination rate constant, estimated by linear regression of logarithmically transformed concentration versus time data.
Terminal phase half life | 48 hours
  Terminal phase half life, estimated using the equation [ln(2)/λz]

CONTACTS AND LOCATIONS:
Overall Officials: Rene Myers, Ph.D., Study Director — scPharmaceuticals, Inc.

IPD SHARING:
Plan to Share IPD: No